CLINICAL TRIAL: NCT05252741
Title: Evaluation Of Levels Of Pigment Epithelium-Derived Factor (PEDF) In Patients With Psoriasis.
Brief Title: Levels of Pigment Epithelium-derived Factor in Patients With Psoriasis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omnia Ahmed Abdelhafez, Resident of Dermatology, Venereology and Andrology Sohag General Hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: soh-Med-22-02-04
Record Dates: First submitted 2022-02-13; First posted 2022-02-23 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: patients with psoriasis (Active Comparator)
  Interventions: Other: serum samples and punch skin biopsies
- Group 2: age-, sex-, BMI-, and weight-matched control subjects. (Placebo Comparator)
  Interventions: Other: serum samples and punch skin biopsies

INTERVENTIONS:
Other: serum samples and punch skin biopsies — we will take serum samples from psoriasis patients and healthy controls and skin punch biopsies from lesional and non-lesional areas in psoriasis patients.

SUMMARY:
Psoriasis is an immune-mediated chronic inflammatory skin disease associated with increase interaction of inflammatory mediators like adipokines. Pigment epithelium-derived factor (PEDF) is one of the most abundant adipokines and have anti-angiogenesis effect. There is a study showed that PEDF level is up-regulated in the sera of psoriasis patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with psoriasis and group of age and sex-matched healthy volunteers will be included as a control group.

Exclusion Criteria:

* Pregnancy.
* Patients with other inflammatory skin disorders.
* Patients on antioxidants or anti-inflammatory drugs.
* Patients on topical or systemic treatment for psoriasis in the last 4 weeks prior to enrollment in the study.
* Patients on systemic retinoids (Acitretin).
* Obesity: body mass index (BMI ) > 30.
* Malignancies e.g squamous cell carcinoma.
* Viral warts.
* Diabetes.
* Hypertension.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
changes in serum and tissue levels of (PEDF) in patients with psoriasis | 12 months
  evaluate serum and tissue level of (PEDF) in patients with psoriasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes